CLINICAL TRIAL: NCT03656627
Title: Safety, Activity, and Pharmacology of Nivolumab in Patients With Advanced Non-Small Cell Lung Cancer and Pre-existing Autoimmune Disease
Brief Title: Nivolumab in Patients With Advanced Non-Small Cell Lung Cancer and Pre-existing Autoimmune Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-42
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Autoimmune Diseases; Non-small Cell Lung Cancer; Rheumatoid Arthritis; Psoriasis; Giant Cell Arteritis; Polymyalgia Rheumatica; Systemic Lupus Erythematosus; Crohn Disease; Multiple Sclerosis; Ulcerative Colitis
Keywords: Autoimmune Diseases; Non-small Cell Lung Cancer; Ulcerative Colitis; Multiple Sclerosis; Crohn Disease; Systemic Lupus Erythematosus; Polymyalgia Rheumatica; Giant Cell Arteritis; Psoriasis; Rheumatoid Arthritis; Nivolumab; Opdivo
MeSH Terms: conditions — Autoimmune Diseases; Carcinoma, Non-Small-Cell Lung; Arthritis, Rheumatoid; Psoriasis; Giant Cell Arteritis; Polymyalgia Rheumatica; Lupus Erythematosus, Systemic; Crohn Disease; Multiple Sclerosis; Colitis, Ulcerative | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab: Autoimmune Diseases Cohort 1 (Experimental): Arms determined by autoimmune type. First cohort consists of patients with:
  Rheumatoid arthritis, psoriasis, giant cell arteritis/polymyalgia rheumatica, systemic lupus erythematosis
  If a patient has more than one autoimmune condition, if all the conditions are within either cohort 1 or 2 above, the patient will be assigned to that cohort. If the patient has conditions from both cohort 1 and 2, the patient will be grouped in cohort 2.
  Interventions: Drug: Nivolumab
- Nivolumab: Autoimmune Diseases Cohort 2 (Experimental): Arms determined by autoimmune type. Second cohort consists of patients with:
  Other autoimmune diseases (ulcerative colitis, Crohn's disease, multiple sclerosis). Patients must be discussed with PI prior to enrollment.
  If a patient has more than one autoimmune condition, if all the conditions are within either cohort 1 or 2 above, the patient will be assigned to that cohort. If the patient has conditions from both cohort 1 and 2, the patient will be grouped in cohort 2.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given as an IV infusion every two weeks, in an outpatient setting. One cycle is a 28-day period, with Nivolumab given on days 1 and 15 of a 28-day cycle.
  For each cohort, all patients will be dosed at 240 mg IV. There will be no dose de-escalation or escalation from this dose level.

SUMMARY:
The purpose of this study is to explore the safety, tolerability and activity of Nivolumab, a PD-1 inhibitor, in cohorts of patients with autoimmune disease. Two cohorts of patients will be enrolled, based on autoimmune disease type.

Patients will be screened within 28 days prior to the start of dosing. Eligible patients will be enrolled in either of the two cohorts. Patients will receive treatment every two weeks, in an outpatient setting. One cycle is a 28-day period, with Nivolumab given on days 1 and 15 of a 28-day cycle. Subjects will be permitted to continue treatment beyond initial RECIST 1.1.

DETAILED DESCRIPTION:
The purpose of this study is to explore the safety, tolerability and activity of Nivolumab, a PD-1 inhibitor, in cohorts of patients with autoimmune disease. Two cohorts of patients will be enrolled, based on autoimmune disease type as outlined below. Entry into cohorts 1 and 2 will start simultaneously and enroll independently.

Cohort 1: Rheumatoid arthritis, psoriasis, giant cell arteritis/polymyalgia rheumatica, systemic lupus erythematosis Cohort 2: Other autoimmune diseases (ulcerative colitis, Crohn's disease, multiple sclerosis). Patients must be discussed with PI prior to enrollment.

Patients will be screened within 28 days prior to the start of dosing. Eligible patients will be enrolled in either of the two cohorts. Patients will receive treatment every two weeks, in an outpatient setting. One cycle is a 28-day period, with Nivolumab given on days 1 and 15 of a 28-day cycle. Subjects will be permitted to continue treatment beyond initial RECIST 1.1. For each cohort, all patients will be dosed at 240 mg IV. There will be no dose de-escalation or escalation from this dose level.

Participants will be followed with telephone follow up for two years after removal from protocol therapy or until death, whichever occurs first. Phone calls will be placed every six months and survival follow up obtained. Participants removed from protocol therapy for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event, in addition to the follow up for two years after removal from protocol therapy or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
3. Metastatic, locally advanced or recurrent NSCLC, not amenable to curative therapy.
4. Patients should have received at least one platinum-based chemotherapy regimen for recurrent or metastatic disease or have received platinum-based chemotherapy as part of adjuvant or neoadjuvant therapy and experienced progression of disease within 6 months of completing therapy.
5. Patients with tumor genetic alterations such as EGFR, ALK, ROS1 or BRAF V600E alterations for which there is FDA-approved targeted therapy must have been treated with the appropriate targeted inhibitors in prior therapy
6. No limit on number of prior therapies
7. Ability to provide written, informed consent
8. Patients must be on a stable regimen of treatment for their autoimmune condition without need for addition of new medications or escalating doses of preexisting medications in the previous 12 weeks prior to study entry
9. In addition, patients with the following autoimmune diseases must have baseline disease activity scores as follows (please see Appendix A):

   * For rheumatoid arthritis: DAS28 < 5.1
   * For polymyalgia rheumatica: PMR-AS < 17
   * For Sjogrens: ESSDAI < 14
   * For ulcerative colitis: SSCAI < 5
   * For Crohn's disease: CDAI < 450
   * For systemic lupus erythroderma: SLEDAI-2K < 20
   * For multiple sclerosis: EDSS < 5.5
10. Adequate organ and marrow function as defined by:

    * absolute neutrophil count ≥ 1,500/mcL
    * platelets ≥ 100,000/mcL
    * total bilirubin ≤ 2.5 × institutional upper limit of normal
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal, OR
    * AST(SGOT)/ALT(SGPT ) ≤5 × institutional upper limit of normal if liver metastases are present
    * Creatinine within normal institutional limits OR
    * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
11. Non-pregnant and non-nursing.
12. Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses > 1 year.
13. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.

Exclusion Criteria:

1. No chemotherapy or radiotherapy within two weeks of study entry. Prior targeted therapy is allowed as long as at least 5 half-lives have elapsed since last dose.
2. All adverse events (other than alopecia) from prior therapy must be resolved to Grade 1 or less.
3. Patients who are known to be HIV positive are excluded due to the known immunologic alterations associated with the disease. HIV testing is not required.
4. No uncontrolled intercurrent illness such as active infection, or psychiatric illness or social situation that in the judgment of the investigator would limit compliance with study requirements
5. No active interstitial lung disease (ILD) or pneumonitis, or a history of ILD or pneumonitis requiring treatment with corticosteroids
6. No live vaccine within 30 days of start of study treatment
7. No carcinomatous meningitis or untreated CNS metastases
8. No history of significant cardiac disease or presence of an abnormality in electrocardiograms that, in the investigator's opinion, is medically exclusionary or clinically meaningful
9. No other active malignancy
10. No known history of or positivity for active hepatitis B or C. HBV DNA and/or HCV RNA must be undetectable and HBsAg must be negative at the time of screening
11. No active unstable angina and/or congestive heart failure, or myocardial infarction within 6 months prior to protocol participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 48 Months
  The DLT determination period is the first six weeks after cycle 1 day 1. Dose limiting toxicities are further defined in the trial protocol.

SECONDARY OUTCOMES:
Overall Response Rate | 48 Months
  Overall response rate is defined to be the best objective status recorded from the start of the treatment until disease progression/recurrence
Progression-Free Survival | 48 Months
  Progression-free survival will be evaluated for each cohort using Kaplan-Meier estimator.
Overall Survival | 48 Months
  Overall survival will be evaluated for each cohort using Kaplan-Meier estimator.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Dartmouth Hitchcock Norris Cotton Cancer Center, Lebanon, New Hampshire
  - The Ohio State University Wexner Medical Center - Thoracic Oncology Clinic, Columbus, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson J, Caplan L, Yazdany J, Robbins ML, Neogi T, Michaud K, Saag KG, O'Dell JR, Kazi S. Rheumatoid arthritis disease activity measures: American College of Rheumatology recommendations for use in clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):640-7. doi: 10.1002/acr.21649. PMID 22473918
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] van der Heijde DM, van Leeuwen MA, van Riel PL, Koster AM, van 't Hof MA, van Rijswijk MH, van de Putte LB. Biannual radiographic assessments of hands and feet in a three-year prospective followup of patients with early rheumatoid arthritis. Arthritis Rheum. 1992 Jan;35(1):26-34. doi: 10.1002/art.1780350105. PMID 1731813
- [Background] Wijnands MJ, van't Hof MA, van Leeuwen MA, van Rijswijk MH, van de Putte LB, van Riel PL. Long-term second-line treatment: a prospective drug survival study. Br J Rheumatol. 1992 Apr;31(4):253-8. doi: 10.1093/rheumatology/31.4.253. PMID 1348198
- [Background] Fransen J, van Riel PL. The Disease Activity Score and the EULAR response criteria. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S93-9. PMID 16273792
- [Background] Leeb BF, Bird HA. A disease activity score for polymyalgia rheumatica. Ann Rheum Dis. 2004 Oct;63(10):1279-83. doi: 10.1136/ard.2003.011379. PMID 15361387
- [Background] Leeb BF, Bird HA, Nesher G, Andel I, Hueber W, Logar D, Montecucco CM, Rovensky J, Sautner J, Sonnenblick M. EULAR response criteria for polymyalgia rheumatica: results of an initiative of the European Collaborating Polymyalgia Rheumatica Group (subcommittee of ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1189-94. doi: 10.1136/ard.2002.002618. PMID 14644857
- [Background] Leeb BF, Rintelen B, Sautner J, Fassl C, Bird HA. The polymyalgia rheumatica activity score in daily use: proposal for a definition of remission. Arthritis Rheum. 2007 Jun 15;57(5):810-5. doi: 10.1002/art.22771. PMID 17530664
- [Background] Seror R, Theander E, Brun JG, Ramos-Casals M, Valim V, Dorner T, Bootsma H, Tzioufas A, Solans-Laque R, Mandl T, Gottenberg JE, Hachulla E, Sivils KL, Ng WF, Fauchais AL, Bombardieri S, Valesini G, Bartoloni E, Saraux A, Tomsic M, Sumida T, Nishiyama S, Caporali R, Kruize AA, Vollenweider C, Ravaud P, Vitali C, Mariette X, Bowman SJ; EULAR Sjogren's Task Force. Validation of EULAR primary Sjogren's syndrome disease activity (ESSDAI) and patient indexes (ESSPRI). Ann Rheum Dis. 2015 May;74(5):859-66. doi: 10.1136/annrheumdis-2013-204615. Epub 2014 Jan 17. PMID 24442883
- [Background] Puzenat E, Bronsard V, Prey S, Gourraud PA, Aractingi S, Bagot M, Cribier B, Joly P, Jullien D, Le Maitre M, Paul C, Richard-Lallemand MA, Ortonne JP, Aubin F. What are the best outcome measures for assessing plaque psoriasis severity? A systematic review of the literature. J Eur Acad Dermatol Venereol. 2010 Apr;24 Suppl 2:10-6. doi: 10.1111/j.1468-3083.2009.03562.x. PMID 20443995
- [Background] Chow C, Simpson MJ, Luger TA, Chubb H, Ellis CN. Comparison of three methods for measuring psoriasis severity in clinical studies (Part 1 of 2): change during therapy in Psoriasis Area and Severity Index, Static Physician's Global Assessment and Lattice System Physician's Global Assessment. J Eur Acad Dermatol Venereol. 2015 Jul;29(7):1406-14. doi: 10.1111/jdv.13132. Epub 2015 Apr 27. PMID 25917315
- [Background] Cooney RM, Warren BF, Altman DG, Abreu MT, Travis SP. Outcome measurement in clinical trials for Ulcerative Colitis: towards standardisation. Trials. 2007 Jun 25;8:17. doi: 10.1186/1745-6215-8-17. PMID 17592647
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] Higgins PD, Schwartz M, Mapili J, Krokos I, Leung J, Zimmermann EM. Patient defined dichotomous end points for remission and clinical improvement in ulcerative colitis. Gut. 2005 Jun;54(6):782-8. doi: 10.1136/gut.2004.056358. PMID 15888785
- [Background] Jowett SL, Seal CJ, Phillips E, Gregory W, Barton JR, Welfare MR. Defining relapse of ulcerative colitis using a symptom-based activity index. Scand J Gastroenterol. 2003 Feb;38(2):164-71. doi: 10.1080/00365520310000654. PMID 12678333
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701
- [Background] Sostegni R, Daperno M, Scaglione N, Lavagna A, Rocca R, Pera A. Review article: Crohn's disease: monitoring disease activity. Aliment Pharmacol Ther. 2003 Jun;17 Suppl 2:11-7. doi: 10.1046/j.1365-2036.17.s2.17.x. PMID 12786607
- [Background] Romero-Diaz J, Isenberg D, Ramsey-Goldman R. Measures of adult systemic lupus erythematosus: updated version of British Isles Lupus Assessment Group (BILAG 2004), European Consensus Lupus Activity Measurements (ECLAM), Systemic Lupus Activity Measure, Revised (SLAM-R), Systemic Lupus Activity Questionnaire for Population Studies (SLAQ), Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), and Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S37-46. doi: 10.1002/acr.20572. No abstract available. PMID 22588757
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Yee CS, Farewell VT, Isenberg DA, Griffiths B, Teh LS, Bruce IN, Ahmad Y, Rahman A, Prabu A, Akil M, McHugh N, Edwards C, D'Cruz D, Khamashta MA, Gordon C. The use of Systemic Lupus Erythematosus Disease Activity Index-2000 to define active disease and minimal clinically meaningful change based on data from a large cohort of systemic lupus erythematosus patients. Rheumatology (Oxford). 2011 May;50(5):982-8. doi: 10.1093/rheumatology/keq376. Epub 2011 Jan 18. PMID 21245073
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237